CLINICAL TRIAL: NCT05867680
Title: A Pilot Feasibility Trial of the Online Mothers and Babies Course (eMB): Improving Perinatal Mental Health for Pregnant Women and Their Partners
Brief Title: Feasibility Trial of an Online Course (eMB) to Reduce Anxiety and Depression for Pregnant Women and Their Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Fahs Beck Fund for Research and Experimentation (Unknown)
Responsible Party: Principal Investigator, Shannon Canfield, Assistant Research Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 000686919
Record Dates: First submitted 2023-04-27; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Anxiety Disorders Generalized; Depression
Keywords: prenatal; Online intervention; randomized control trial; feasibility; couples; Cognitive Behavioral Therapy
MeSH Terms: conditions — Generalized Anxiety Disorder; Depression

STUDY DESIGN:
Intervention Model Description: Random assignment to the control or treatment group using a 1:1 parallel assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Treatment group participants received the eMB intervention during the 8-week trial period.
  Interventions: Behavioral: Online Mothers and Babies Course (eMB)
- Control (No Intervention): The control group received a PDF community resources informational sheet, also available to the intervention group via the eMB program.

INTERVENTIONS:
Behavioral: Online Mothers and Babies Course (eMB) — The eMB is an online, asynchronous, self-administered intervention modeled after the efficacious and in-person Mothers and Babies Course. (4) The eight-week course includes psychoeducational modules containing YouTube videos, vignettes, interactive quizzes, homework, guided meditations, and downloadable resources that teach strategies to promote a healthy outcome for mothers and their newborns: 1) overview, 2) thoughts and my mood, 3) fighting harmful and increasing helpful thoughts, 4) activities and my mood, 5) pleasant activities help make a healthy reality, 6) contact with others and my mood, 7) planning for the future and graduation, 8) relaxation exercises.
  Arms: Treatment

SUMMARY:
This pilot study engaged pregnant couples experiencing elevated symptoms of maternal anxiety or depression with an existing online psychoeducation intervention, the Online Mothers and Babies Course (eMB). The study had three primary aims to assess overall feasibility; 1) explore the feasibility of delivering eMB to couples by assessing recruitment, retainment, and adherence, 2) examine eMB's preliminary efficacy for reducing PMAD symptoms, and 3) describe participants' satisfaction and perceptions about eMB acceptability.

The intervention group received the 8-week eMB and the control group received an informational resources sheet.

DETAILED DESCRIPTION:
Perinatal anxiety and depression are common, often co-morbid, and occur more frequently than outside pregnancy. Preventative measures can reduce the risk of poor mental and physical health outcomes and improve coping self-efficacy and the perception of social support. The antenatal period is an optimal time for intervention. Efficacious interventions include engaging pregnant people in cognitive-behavioral therapy and increasing the pregnant person's perception of social support -particularly partner support. Despite the evidence that partners can buffer stressors and, more generally, that perceived social support is protective, there are few interventions to reduce symptoms of anxiety or depression that involve partners. Online interventions can effectively manage mental health, increase knowledge and access to resources, and improve social connectivity. Online interventions have decreased perinatal anxiety, depression, and perception of stress, increased awareness about mental health risk factors and protective strategies, and improved coping self-efficacy successfully. Although perceived partner support is protective against poor mental health for pregnant people, partners' potential roles in online interventions is an understudied area of intervention innovation. Expanding the number of effective and equitably accessible online interventions is essential, given structural and social barriers to care.

Engaging the pregnant person and her partner as a dyad in perinatal studies complicates recruitment, retention, adherence, and longitudinally measuring change. This pilot study engaged pregnant couples experiencing elevated symptoms of maternal anxiety or depression with an existing online psychoeducation intervention, the Online Mothers and Babies Course (eMB). The study had three primary aims to assess overall feasibility; 1) explore the feasibility of delivering eMB to couples by assessing recruitment, retainment, and adherence, 2) examine eMB's preliminary efficacy for reducing PMAD symptoms, and 3) describe participants' satisfaction and perceptions about eMB acceptability.

Analytic Approach The approach follows Whitehead et al. (2016) guidance on sample size to complete a pilot feasibility trial; a sample size of 30 people for each condition was necessary. (1) The study uses univariate analysis to calculate descriptive statistics describing the sample and feasibility outcomes.

Given the study's aims, the study hypothesized that it would be feasible to deliver the program to pregnant couples and there would be a significant reduction in anxiety and depression symptoms in favor of the intervention group. A factorial Analysis of Variance (ANOVA) with repeated measures on the dyadic role and survey time was used to test the study hypotheses. The analysis used an intention-to-treat analysis approach and a significance level of α = 0.05 or less. Repeated measures were recorded three times for each participant and each outcome of interest to evaluate the effect of the eMB course. Based on the minimum Akaike Information Criterion (AIC), researchers used an optimal residual covariance structure for each outcome. When factor interactions were significant, posthoc comparisons were used. The study retained data when available and dropped cases missing at times two or three. Data missing in this study are considered missing at random and analyzed with maximum likelihood estimation. Analyses were conducted using SPSS software.

To assess the degree of program satisfaction, item responses were summed, and the average satisfaction score was calculated for the intervention group. Interview data were analyzed using an inductive thematic approach. Both authors are PhD-trained researchers with extensive qualitative experience and contributions to various health and social science studies. The analysis occurred in stages: preparing transcripts after Zoom download, becoming familiar with the data, creating memos, coding (i.e., applying labels to text segments), searching for patterns in the coding, defining and naming themes from patterns, and writing up results. Analysis was conducted in Dedoose. The study investigator completed each stage first, and a member check was conducted by the second researcher.

ELIGIBILITY:
Inclusion criteria:

* Adult, cis-gender and heterosexual pregnant people
* Pregnancy between 13- and 30 weeks gestation
* Elevated symptoms of pregnancy anxiety or depression (i.e., above the cut-off of 10 with validated measures - the Patient Health Questionaire-9 (PHQ-9; 33) or the Generalized Anxiety Disorder-7 (GAD-7; 29)
* Enrolled as a couple with the pregnant person and their partner cohabitating in Missouri and having internet access

Exclusion criteria:

* If either person in the couple did not meet the inclusion criteria
* Endorsed suicide risk,
* Could not comprehend the consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender women; cisgender men
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | Change between baseline, week 4 and 8
  The GAD-7 has seven self-reported items assessing general anxiety levels and has good reliability (α =.89). The responses are scored zero to three based on symptom severity, and the sum of all items ranges from zero to 21. A score of five, 10, and 15 are cut points for mild, moderate, and severe anxiety. (Spitzer et al.2006)
Edinburgh Postnatal Depression Scale (EPDS) | Change between baseline, week 4 and 8
  The EPDS is a ten-item self-reported questionnaire validated for use in pregnancy, acceptable for use with partners, and found to have good reliability (α = .87). The item responses are scored from zero to three to indicate symptom severity, and three questions are reverse-scored. A total score ranges from zero to 30. A score of ten or more indicates moderate symptom severity and is considered the optimal cut-off for further assessment or intervention.(Murry and Cox, 1990)
Implementation feasibility | Upon trial completion
  For feasibility measures, we used study tracking data and Qualtrics usage analytics; these include recruitment, retention and attrition rates, and participant intervention adherence. The recruitment rate is the proportion of study inquiries and enrollments. Retention is the portion of survey completions and the reminders at each measurement time for each person. Attrition is the proportion of enrolled dyads and dropouts (i.e., both members failed to complete the final two surveys).
Intervention adherence | Upon trial completion
  Intervention adherence is the average number of participants completing one lesson per week, the proportion of fully or partially complete lessons, and the average total lessons visited. An additional descriptive usage measure was captured with a multiple-option survey item asking whether the participant used eMB alone, together with their counterparts, a combination of alone and together, or not at all.
Client Satisfaction Questionnaire (CSQ-8) | week 8
  The CSQ-8 is a 4-point Likert scale with responses ranging from strongly disagree to agree strongly and is sum-scored from eight to 32. A score from eight to 13 is interpreted as "poor," 14-19 as "fair," 20-25 as "good," and 26-32 as "excellent" satisfaction. The scale has high internal consistency (α = .9) and is used routinely in healthcare research (Attkisson & Greenfield, 1995). Satisfaction and program acceptability are also measured qualitatively using semi-structured interviews. Questions included prompts about the helpfulness of materials, ease of use, areas for improvement, and how the course improved coping behaviors.(Attkisson & Zwick, 1982)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] R. F. Muñoz, H.-N. Le, C. G. Ippen, M. A. Diaz, G. G. Urizar Jr, J. Soto, et al. Cognitive and Behavioral Practice 2007 Vol. 14 Issue 1 Pages 70-83
- [Background] Moran TE, O'Hara MW. A partner-rating scale of postpartum depression: the Edinburgh Postnatal Depression Scale - Partner (EPDS-P). Arch Womens Ment Health. 2006 Jul;9(4):173-80. doi: 10.1007/s00737-006-0136-x. Epub 2006 Jun 8. PMID 16755331
- [Background] Murray D, Cox JL. Screening for depression during pregnancy with the Edinburgh Depression Scale (EDDS). J Reprod Infant Psyc. 1990;8(2):99-107.
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Derived] Canfield SM, Canada KE, Rolbiecki AJ, Petroski GF. Feasibility and acceptability of an online mental health intervention for pregnant women and their partners: a mixed method study with a pilot randomized control trial. BMC Pregnancy Childbirth. 2023 Oct 18;23(1):739. doi: 10.1186/s12884-023-06031-4. PMID 37853333